CLINICAL TRIAL: NCT01213134
Title: Evaluating the Implementation of Portfolio Assessment in Resident Training Program
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Wei-Pin Ho, Department of Orthopaedics
Other Study IDs: 98TMU-WFH-13
Record Dates: First submitted 2010-09-30; First posted 2010-10-01 (Estimated); Last update posted 2010-10-01 (Estimated); Status verified 2010-09

CONDITIONS: Residents' Perceptions on Portfolio Use in Clinical Training
Keywords: Medical Education; Resident Training; Portfolio

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Portfolios are the records of learning process, providing evidences of experiential learning. It can be a valuable tool not only for understanding the learning process but also for evaluating the accomplishment. Portfolios promote learners to reflecting, thinking, improving in learning as well as achieving learning goals. It has been widely applied in medical education. The goals of resident training outcomes in Wan-Fang Hospital are the ACGME six core competences. The Wan-Fang hospital, one of Taipei Medical University affiliated hospitals and the first implementing portfolio assessment teaching hospitals in Taiwan, will conduct portfolio assessment to assess residents competences. Facilitating residents bring reflective learning into practice, personal and professional growth and demonstrating the outcomes of training program. This study describes initiating and implementing portfolio assessment procedures. Qualitative and quantitative research methods are applied for evaluating the portfolio assessment process and the data of validity and reliability. Qualitative data collection methods of interview, focus groups and meetings will be used understanding the experiences and viewpoints of residents, mentors and assessors. Then quantitative data collection method of questionnaire will be subsequently used. The results of this study will provide experiences and suggestions for the implementation of portfolio assessment system in medical education.

ELIGIBILITY:
Inclusion Criteria:

* residents in Wanfang Hospital willing to be enrolled to this study

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: residents tutors
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-05 (Estimated); Study Completion 2012-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Pin Ho, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan